CLINICAL TRIAL: NCT03274505
Title: Comparison of the Prevalence of Sleep Disorders in Transient Ischemic Attack and Stroke
Brief Title: Sleep Disorders in Transient Ischemic Attack and Stroke: SOMN'AIC Study
Acronym: SOMN'AIC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0418
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Sleep Disorder; Stroke
MeSH Terms: conditions — Sleep Wake Disorders; Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: Patients seen by a rehabilitation physician at a routine 3 months' post-stroke examination
  Interventions: Other: Questionnaires
- TIA patients: Patients seen by a stroke specialist at the "SOS TIA" examination
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — * Questionnaires about excessive daytime sleepiness (Epworth scale), insomnia (Severity of Insomnia Scale), Restless Legs Syndrome, Chronotype (Horne and Ostberg questionnaire), Sleep apnoea syndrome (Berlin questionnaire)
  * Clinical evaluation
  * Routine neuropsychological evaluation (for stroke patients)
  * Routine Polysomnography for patients with high suspicion of sleep apnoea syndrome (SOS score (Epworth + Berlin) > 10)

SUMMARY:
Sleep disorders in the setting of stroke are numerous, including sleep-related breathing disorders, insomnia, excessive daytime sleepiness and restless legs syndrome. Consequences of theses sleep disturbances include impaired functional outcome and quality of life, anxious and depressive troubles and increased cardio-vascular morbi-mortality. Mechanisms underlying sleep disorders in the setting of stroke are complex and still partly elucidated. They probably involve the consequences of the ischemic lesion and of the handicap, but also of associated vascular risk factors and more generally pre-existent medical history, or they could represent themselves a risk factor for stroke. Transient ischemic attack (TIA) is a particular condition in which risk factors and background of patients are similar to that observed in stroke, without any cerebral lesion and no persistent neurological deficit. The main objective of the SOMN'AIC study is to compare the prevalence of sleep disorders in stroke and in transient ischemic attack (TIA). The study hypothesis is that the prevalence of sleep disorders may be higher in stroke than in TIA patients, reflecting the consequences of the lesion and the associated handicap.

ELIGIBILITY:
Inclusion Criteria:

* Stroke group: patients with a diagnosis of stoke and seen at the routine post-stroke 3 month' rehabilitation examination
* TIA group: diagnosis of a TIA by a stroke specialist at the "SOS TIA" examination
* > 18 years

Exclusion Criteria:

* Refusal to participate
* Severe cognitive impairment leading to inability to fulfil questionnaires
* For the TIA group: presence of an ischemic lesion on CT scan or MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke and transient ischemic attack patients
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Comparison of stroke and transient ischemic attack population regarding the prevalence of the presence of at least one sleep disorder | Maximum 9 months
  Presence of at least one of the following sleep disorders assessed by clinical evaluation, questionnaires +/- polysomnography: insomnia, excessive daytime sleepiness (EDS), restless legs syndrome (RLS) and sleep apnoea syndrome (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Laure PETER-DEREX, MD, PhD, Principal Investigator — Centre de Médecine du Sommeil et des Maladies respiratoires, CH de la Croix Rousse - HCL
Locations (3):
- France (3):
  - Service de Neurologie Vasculaire Groupement Hospitalier Est, Bron
  - Sleep Medicine Center, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon
  - Service de MPR- Hôpital Henry Gabrielle - Groupement Sud, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No